CLINICAL TRIAL: NCT02348099
Title: Ultrasound Guided Detection and Characterization of Subclinical Lipohypertrophy in Type 1 and Type 2 Diabetes Mellitus
Brief Title: Ultrasound Detection and Characterization of Subclinical Hypertrophy in Diabetes
Status: Terminated | Type: Observational
Why Stopped: The study run its course
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Graydon Meneilly, Professor, UBC Department of Medicine, University of British Columbia
Other Study IDs: H14-02461
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Results first posted 2025-04-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Lipohypertrophy
Keywords: Diabetes; Lipohypertrophy; Ultrasound
MeSH Terms: conditions — Diabetes Mellitus | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound — Abdomen scanned with portable ultrasound to determine presence of subclinical lipohypertrophy.

SUMMARY:
This is a pilot study to enroll 100 people to assess the incidence of lipohypertrophy as detected with ultrasound and its impact on glycemic variability.

DETAILED DESCRIPTION:
Lipohypertrophy is a well documented phenomenon in patients with diabetes in which hypertrophy and differentiation of adipocytes occurs in the dermal reticular layer at the sites of subcutaneous insulin injection. Currently, lipohypertrophy is assessed by palpating insulin injection sites. The detection on early, non palpable (subclinical) lipohypertrophy remains difficult in the clinical setting. Recent studies have identified distinct ultrasonographic features of hyperechogenicity in areas of adipose tissue consistent with clinical evidence of lipohypertrophy at insulin injection sites, and have detected changes int he thickness of subcutaneous tissue where not clinically evident in population of patients with type 1 diabetes. Lipohypertrophy can adversely affect glycemic control. Injecting into lipohypertrophic areas leads to poor absorption and the need for increasing doses of insulin.

In this study study participants will undergo an assessment for lipohypertrophy during a scheduled visit at the VGH Diabetes Centre. A Diabetes Nurse will assess lipohypertrophy by palpation according to the FIT Protocol. A second diabetes nurse who was not present at the palpation will assess insulin injection sites for lipohypertrophy by ultrasound using a linear probe.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Type 1 or Type 2 diabetes
* Using insulin to manage diabetes for at least 2 years

Exclusion Criteria:

* Using insulin pumps, insulin secretagogues, Glucagon-Like Peptide-1 (GLP-1) agonists to manage diabetes
* Use of immunosuppressant agents
* Women who are pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People age 19 and over with type 1 or type 2 diabetes who take insulin to manage their diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graydon Meneilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapeluto JE, Paty BW, Chang SD, Meneilly GS. Ultrasound detection of insulin-induced lipohypertrophy in Type 1 and Type 2 diabetes. Diabet Med. 2018 Oct;35(10):1383-1390. doi: 10.1111/dme.13764. Epub 2018 Jul 16. PMID 29908078

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetes Patients Treated With Insulin: We propose a pilot study in a minimum of 100 patients with diabetes who have been using insulin therapy for at least two years and being treated with insulin at the time of the study. Patients using insulin pumps, insulin secretagogues (e.g. sulfonylureas), GLP-1 agonists and immunosuppreressant agents will be excluded. Women who are pregnant will be excluded.
Period: Overall Study
Arm/Group | Diabetes Patients Treated With Insulin
Started | 100
Completed | 100 (This study is consisted in one Phase. During this Phase we have determined the percentage of patients who have subclinical lipohypertrophy in Phase 1 will be offered enrollment to assess glycemic correlation in areas of subclinical lipohypertrophy.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This is a pilot study in a minimum of 100 patients with diabetes who have been using insulin therapy for at least two years and being treated with insulin at the time of the study.
Arm/Group | Diabetes Patients Treated With Insulin
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 20
Age, Continuous [Mean (Full Range); unit: years] | 50 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 30
  More than one race | 15
  Unknown or Not Reported | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 100
Presence of Lipohypertrophy [Number; unit: participants] | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of Subclinical Lipohypertrophy
Description: Lipohypertrophy seen on ultrasound but not felt by palpation
Time Frame: Assessed one time only at the time of clinic visit
Population: 100 participants were analyzed for having subclinical lipohypertophy.
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetes Patients Treated With Insulin
Number analyzed (Participants) | 100
Participants | 20
Statistical Analysis 1: Comparison: Diabetes Patients Treated With Insulin; A student's paired t-test will be used to determine the difference if any in CV of glucose between injection sited. If the null hypothesis is true, it suggests that any changes witnessed in an experiment are because of random chance and not because of changes made to variables in the experiment. A "power calculation" is a statistical method used to determine the minimum sample size needed to detect a statistically significant effect of a certain size; Test type: Other — A student's paired t-test will be used to determine the difference if any in CV of Glucose between injection sites. In the third phase, area under the curve will be measured to determine differences between insulin absorption levels. Statistical analysis will be performed using SPSS version 15.0.0 and SAS version 8.2 A "power calculation" is a statistical method used to determine the minimum sample size needed to detect a statistically significant effect of a certain size; p < 0.01, t-test, 2 sided; Odds Ratio (OR) = 95; a P-Value is <0.01

ADVERSE EVENTS:
Time Frame: During study procedure within study visit up to 1 hour
Description: All adverse events will be collected from the enrolled participants by the study staff
Groups:
- Diabetes Patients Treated With Insulin: We propose a pilot study in a minimum of 100 patients with diabetes who have been using insulin therapy for at least two years and being treated with insulin at the time of the study. Patients using insulin pumps, insulin secretagogues (e.g. sulfonylureas), GLP-1 agonists and immunosuppreressant agents will be excluded. Women who are pregnant will be excluded.
  There may be some discomfort associated with the insertion of the glucose sensor. There is a small risk of skin infection from the insertion of the glucose sensor and catheter and the possibility of an allergic reaction from the tape used to apply it. This risk occurs less than 1 in 1000 times the sensor is used. If patients have concerns regarding insulin dose adjustments they will have access to a diabetes education and research nurse who can assist with insulin dose titration. Any additional adverse events will be monitored by a trained research nurse at the Diabetes Centre.
Arm/Group | Diabetes Patients Treated With Insulin
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 1/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Patients Treated With Insulin (N=100)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) — Skin infection from the insertion of the glucose sensor and catheter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02348099/Prot_SAP_000.pdf